CLINICAL TRIAL: NCT06271447
Title: Answerability and Minimal Clinical Significance of the Turkish Versions of the Fear-Avoidance Beliefs Questionnaire, Tampa Kinesiophobia Scale, and Pain Catastrophizing Scales in Patients With Non-Specific Chronic Low Back Pain
Brief Title: Answerability and Minimal Clinical Significance of the Pain Questionnaires
Status: Recruiting | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-21-705
Record Dates: First submitted 2024-02-14; First posted 2024-02-21 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Chronic Low-back Pain
Keywords: Chronic Low Back Pain; pain management; rehabilitation; minimal clinical significance
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Other: Traditional therapy — All participants will receive a 60-minute individual treatment program consisting of 16 sessions of routine physiotherapy aimed at reducing pain and improving function over four weeks. These treatments are already the patient's routine physiotherapy modalities. No changes will be made to the study.
  Since the questionnaires to be used in the study are related to fear of movement and pain, neuroscience education will be included in the treatment program of the patients. Patients will be informed about proper posture and movement regarding fear of movement and pain avoidance behaviors.

SUMMARY:
To investigate the reliability and sensitivity of the Turkish versions of the Fear-Avoidance Beliefs Questionnaire, Tampa Scale for Kinesiophobia, and The Pain Catastrophizing Scale in patients with chronic non-specific low back pain undergoing multidisciplinary rehabilitation.

DETAILED DESCRIPTION:
Nonspecific chronic low back pain is a common condition that can have a significant impact on patient's daily lives and beliefs. Patients often believe that there is a strong relationship between structural changes in the lower back, pain, and activities of daily living. Patients with nonspecific low back pain may have lower expectations for recovery because they tend to believe that their condition is chronic and unlikely to improve significantly. Patients' beliefs and perceptions of their condition can influence the clinical management of low back pain. Tampa Scale for Kinesiophobia (TSK), Fear-Avoidance Beliefs Questionnaire (FABQ), and The Pain Catastrophizing Scale (PCS) are commonly used in patients with non-specific chronic low back pain. The common feature of these scales is that they evaluate issues such as pain perception, pain-related beliefs, and pain coping strategies. The use of these scales can provide important information to better respond to individuals' needs in pain management and rehabilitation processes. However, the minimal clinical relevance and answerability of the surveys were not explicitly discussed in the search results. Further research is needed to investigate the clinical consequences of fear-avoidance beliefs and their potential impact on treatment outcomes for patients with chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Getting diagnosed with chronic non-specific low back pain
* Being able to read and speak Turkish
* Being between the ages of 18 and 65
* Agreeing to participate in the research and signing the voluntary consent form.

Exclusion Criteria:

* Presence of systemic disease
* Cognitive impairment status (Mini-Mental State Examination <24),
* Recent (<12 weeks) history of myocardial infarction, cerebrovascular accident
* Presence of radiculopathy, infection, tumor, osteoporosis, vertebral fracture, trauma and surgery in the lumbar region
* Having previously received any exercise therapy and/or training in pain neuroscience.
* Refusal of treatment or failure to comply with treatment

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 100 patients diagnosed with chronic nonspecific low back pain (documented history of low back pain lasting more than twelve weeks without a recognizable, specific pathoanatomical cause of the pain) who applied to the Physical Therapy and Rehabilitation Polyclinic of the hospitals in the Acıbadem Health Group and the Physiotherapy and Rehabilitation Department of Avicenna Ataşehir Hospital will be included in the study. Diagnoses will be given by Health Physical Medicine and Rehabilitation Doctors with at least 20 years of experience. At the first meeting, eligible participants will be informed about the study, potential participants will be screened in terms of inclusion criteria, and verbal and written informed consent will be obtained from eligible participants by the Helsinki criteria.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | baseline and through study completion, an average of 4 weeks
  Visual Analog Scale (VAS) is a pain rating scale used in clinical and research settings to measure the intensity or frequency of various symptoms. In the current study, VAS will be used to record participants' pain intensity. VAS consists of a single 10 cm line; The left end is described as "No pain" and the right end is described as "The most severe pain ever experienced". Patients will be asked to mark the severity of their current pain on a 10 cm line. When calculating, the marked point will be measured in cm. An increase in the score means that the intensity of the pain increases.
Fear-Avoidance Beliefs Questionnaire | baseline and through study completion, an average of 4 weeks
  Fear-Avoidance Beliefs Questionnaire is a tool used to assess fear-avoidance beliefs in patients with low back pain. In the current study, the fear and avoidance behaviors of the participants will be evaluated with FABQ. In the survey, which consists of sixteen questions and two subscales (physical activity and work), each question is scored on a six-point Likert scale (0: strongly disagree; 5: strongly agree). A high score in the evaluation is considered to indicate an increase in fear-avoidance behavior.
Tampa Scale for Kinesiophobia | baseline and through study completion, an average of 4 weeks
  The Tampa Scale for Kinesiophobia (TSK) will be used to assess participants' fear of movement. TSK is a 17-item scale developed to describe the fear of movement or re-injury. Each question is scored on a four-point Likert scale (1: strongly disagree; 4: strongly agree). The scoring of four items was reversed (items 4, 8, 12, and 16). Higher scores represent an increased fear of movement.
The Pain Catastrophizing Scale | baseline and through study completion, an average of 4 weeks
  The Pain Catastrophizing Scale will be used to assess participants' pain-related thoughts and feelings. It is self-administered and consists of 13 items and 3 subscales (helplessness, magnification, and rumination). It is scored using a five-point Likert-type scale (0: never; 4: always). High scores indicate high levels of catastrophizing.
The Perceived Global Impact | through study completion, an average of 4 weeks
  The Global Perceived Impact Scale (GAES) is the usual gold standard for assessing minimal clinically significant change associated with pain in a patient's subjective perception of improvement (global perceived impact). In the current study, the amount of improvement in symptoms perceived by the participants will be evaluated at the end of treatment with GAES. Participants were asked "How would you describe your current condition compared to the beginning of treatment?" question will be asked. They will be asked to rate on a seven-point Likert scale (1: no change or things have gotten worse; 7: much better, a significant improvement). A score of 6 or above will be chosen as the threshold for clinically significant improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Elif E Safran, asst. prof., Principal Investigator — Acibadem University; Irmak I Çavuşoğlu, asst. prof., Study Chair — Acibadem University; Nuray N Alaca, assoc. prof., Study Director — Acibadem University
Locations (1):
- Elif Esma Safran, Istanbul, None Selected, Turkey (Türkiye)